CLINICAL TRIAL: NCT02847286
Title: AN OPEN-LABEL, RANDOMISED TRIAL, WITH A THREE-PERIOD CROSSOVER PART IN HEALTHY HIV-NEGATIVE WOMEN TO ASSESS THE DRUG-DRUG INTERACTION POTENTIAL BETWEEN DAPIVIRINE VAGINAL RING-004, CONTAINING 25 MG OF DAPIVIRINE, AND CLOTRIMAZOLE 10 mg/g (1%) ADMINISTERED AS A VAGINAL CREAM, WITH A FOLLOW-ON PERIOD TO ASSESS THE EFFECT OF MULTIPLE RING REMOVALS AND RE-INSERTIONS DURING THE 28-DAY PERIOD OF THE DAPIVIRINE VAGINAL RING-004 USE ON THE SYSTEMIC AND LOCAL EXPOSURE AND RESIDUAL AMOUNT OF DAPIVIRINE IN USED RINGS
Brief Title: To Assess the Drug-drug Interaction Potential Between Dapivirine Vaginal Ring-004, Containing 25 mg of Dapivirine, and Clotrimazole 10 mg/g (1%)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IPM 036
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: HIV- Prevention
MeSH Terms: interventions — Clotrimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment A (Active Comparator): Dapivirine Ring-004 for 28 days
  Interventions: Drug: Dapivirine Ring-004
- Treatment B (Active Comparator): Dapivirine Ring-004 for 28 days along with clotrimazole, 5 g per day for 7 days
  Interventions: Drug: Dapivirine Ring-004 for 28 days along with clotrimazole
- Treatment C (Active Comparator): Clotrimazole, 5 g per day for 7 days
  Interventions: Drug: Clotrimazole

INTERVENTIONS:
Drug: Dapivirine Ring-004 — Treatment A: Dapivirine Ring-004 for 28 days
  Other Names: Treatment A
  Arms: Treatment A
Drug: Dapivirine Ring-004 for 28 days along with clotrimazole — Treatment B: Dapivirine Ring-004 for 28 days along with clotrimazole, 5 g per day for 7 days
  Other Names: Treatment B
  Arms: Treatment B
Drug: Clotrimazole — Treatment C: Clotrimazole, 5 g per day for 7 days
  Other Names: Treatment C
  Arms: Treatment C

SUMMARY:
A Study to assess the drug-drug interaction potential, between Dapivirine Vaginal Ring-004, containing 25 MG of Dapivirine.

DETAILED DESCRIPTION:
AN OPEN-LABEL, RANDOMISED TRIAL, WITH A THREE-PERIOD CROSSOVER PART IN HEALTHY HIV-NEGATIVE WOMEN TO ASSESS THE DRUG-DRUG INTERACTION POTENTIAL BETWEEN DAPIVIRINE VAGINAL RING-004, CONTAINING 25 MG OF DAPIVIRINE, AND CLOTRIMAZOLE 10 mg/g (1%) ADMINISTERED AS A VAGINAL CREAM, WITH A FOLLOW-ON PERIOD TO ASSESS THE EFFECT OF MULTIPLE RING REMOVALS AND RE-INSERTIONS DURING THE 28-DAY PERIOD OF THE DAPIVIRINE VAGINAL RING-004 USE ON THE SYSTEMIC AND LOCAL EXPOSURE AND RESIDUAL AMOUNT OF DAPIVIRINE IN USED RINGS

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible to enrol in the trial:

1. Women 18 and ≤ 45 years of age who can give written informed consent
2. Available for all visits and consent to follow all procedures scheduled for the trial
3. Healthy, based on medical history, vital signs, physical examination, urinalysis (dipstick and microscopy), laboratory evaluations for genital infections (bacterial vaginosis, gonorrhoea, chlamydia and trichomonas), and laboratory evaluations for haematology and chemistry
4. HIV-negative as determined by an HIV test at the time of screening
5. On a stable form of contraception, defined as:

A stable oral contraceptive regimen for at least 2 months prior to enrolment, OR Transdermal contraceptive patch for at least 3 months prior to enrolment, OR Long-acting progestins for at least 6 months prior to enrolment, OR An intra-uterine device (IUD) inserted (with no vaginal or gynaecological complaints associated with its use) at least 3 months prior to enrolment, OR Have undergone surgical sterilisation at least 3 months prior to enrolment, AND willing to use oral contraceptives if necessary to delay menstruation during the vaginal sampling period 6. Upon pelvic examination at the time of enrolment, the cervix and vagina appear normal as determined by the Investigator/Physician Asymptomatic for genital infections at the time of enrolment (if a woman is diagnosed with any treatable STI, either clinically or by laboratory test at the time of screening, she must complete treatment prior to enrolment) 8. Willing to refrain from the use of topical vaginal medications, vaginal products or objects, including female condoms, tampons, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method), douches, lubricants, vibrators/dildos, and drying agents for 14 days prior to enrolment and for the duration of the trial 9. Documentation of no abnormality on cervical cytology, including grossly bloody smear, within 90 days prior to screening 10. Willing to refrain from participation in any other research trial for the duration of this trial 11. Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures, e.g. by home visit or telephone, or via family or close neighbour contacts (confidentiality to be maintained) 12. Willing to agree to abstain for a total of 2 days (48 hours) prior to each trial visit from: Penile-vaginal intercourse Oral contact with her genitalia 13. Hepatitis B and C negative at the time of screening

Exclusion Criteria:

Participants who have any of the following criteria are NOT eligible to enrol in the trial:

1. Currently pregnant or had their last pregnancy outcome within 3 months prior to screening
2. Currently breast-feeding
3. Currently or within 2 months of participation in any other clinical research trial involving investigational or marketed products prior to screening
4. Untreated symptomatic urogenital infections, e.g. urinary tract or other STIs, or other gynaecological conditions such as vaginal itching, pain, or discharge within 14 days prior to enrolment
5. History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction, incontinence, urge incontinence or an anatomical variation that will not allow placement or retention of the ring
6. Current vulvar or vaginal symptoms/abnormalities that could influence the trial results
7. Cervical cytology at screening that requires cryotherapy, biopsy, treatment (other than for infection), or further evaluation
8. Symptomatic genital herpes simplex virus (HSV) infection or a history of genital herpetic infection
9. Any Grade 2, 3 or 4 haematology, biochemistry or urinalysis laboratory abnormality at baseline (screening) according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events; Addendum 1 Female Genital Grading Table for Use in Microbicide Studies
10. Unexplained, abnormal bleeding per vagina during or following vaginal intercourse, or gynaecologic surgery within 90 days prior to enrolment
11. Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex or silicone
12. Any serious acute, chronic or progressive disease (e.g. any known history of neoplasm, cancer, diabetes, epilepsy, cardiac disease, autoimmune disease, HIV, Acquired Immunodeficiency Syndrome [AIDS], or blood dyscrasias), or signs of cardiac disease, renal failure, or severe malnutrition
13. Have undergone a hysterectomy
14. Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives.

    Participants who have the following criterion are NOT eligible for Treatment F:
15. Using a hormonal intrauterine device.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

PRIMARY OUTCOMES:
Dapivirine concentrations in plasma | 28-day
  Dapivirine concentrations in plasma, measured at specified time points during each 28-day period that the ring is inserted, and for 14 days following ring removal
Clotrimazole concentrations in plasma | 7 days of once daily dosing, and for 14 days after the last administration
  Clotrimazole concentrations in plasma, measured at specified time points during 7 days of once daily dosing, and for 14 days after the last administration.

SECONDARY OUTCOMES:
Dapivirine concentrations in vaginal fluid | 28 days
  Dapivirine concentrations in vaginal fluid, collected at the cervix, measured at specified time points during each 28-day period that the ring is inserted, and for three days following ring removal.
Clotrimazole concentrations in vaginal fluid | 7 days of once daily dosing, and following 14 days after the last administration.
  Clotrimazole concentrations in vaginal fluid, measured at specified time points during 7 days of once daily dosing, and following 14 days after the last administration.

IPD SHARING:
Plan to Share IPD: No